CLINICAL TRIAL: NCT03059355
Title: A Phase I/II, Randomized, Placebo-controlled Comparative Study to Evaluate the Safety and Potential Efficacy of Intravenous Infusion of Umbilical Cord Tissue (UC) Derived Mesenchymal Stem Cells (MSCs) Versus Bone Marrow (BM) Derived MSCs to Evaluate Cytokine Suppression in Patients With Chronic Inflammation Due to Metabolic Syndrome.
Brief Title: Infusion of Umbilical Cord Versus Bone Marrow Derived Mesenchymal Stem Cells to Evaluate Cytokine Suppression.
Acronym: CERES
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID-19 Pandemic and lack of funding
Sponsor: Joshua M Hare (Other)
Collaborators: The Marcus Foundation (Other)
Responsible Party: Sponsor-Investigator, Joshua M Hare, Director of ISCI, Louis Lemberg Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20170095
Record Dates: First submitted 2017-02-06; First posted 2017-02-23 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Endothelial Dysfunction; Metabolic Syndrome; Chronic Inflammation
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pilot phase is open-label. Randomized phase is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Pilot Phase: Group 1 (UCMSCs - 20 million) (Experimental): Three (3) subjects will be treated with a single administration of 2 x 10^7 (20 million) UCMSCs delivered via peripheral intravenous infusion.
  Interventions: Biological: UCMSCs
- Pilot Phase: Group 3 (UCMSCs - 100 million) (Experimental): Three (3) subjects will be treated with a single IV administration of 1 x 10^8 (100 million) UCMSCs delivered via peripheral intravenous infusion.
  Interventions: Biological: UCMSCs
- Pilot Phase: Group 2 (BMMSCs - 20 million) (Experimental): Three (3) subjects will be treated with a single IV administration of 2 x 10^7 (20 million) BMMSCs delivered via peripheral intravenous infusion.
  Interventions: Biological: BMMSCs
- Pilot Phase: Group 4 (BMMSCs -100 million) (Experimental): Three (3) subjects will be treated with a single IV administration of 1 x 10^8 (100 million) BMMSCs delivered via peripheral intravenous infusion.
  Interventions: Biological: BMMSCs
- Group A (UCMSCs - 100 million) (Experimental): Participants randomized to receive a single administration of 1 x 10^8 (100 million) UCMSCs delivered via peripheral intravenous infusion.
  Interventions: Biological: UCMSCs
- Group B (BMMSCs - 100 million) (Experimental): Participants randomized to receive a single administration of 1 x 10^8 (100 million) BMMSC delivered via peripheral intravenous infusion.
  Interventions: Biological: BMMSCs
- Group C (Placebo) (Placebo Comparator): Participants randomized to receive a single administration of placebo via peripheral intravenous infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: UCMSCs — Allogeneic Umbilical Cord Tissue derived MSCs (UCMSCs)
  Arms: Group A (UCMSCs - 100 million); Pilot Phase: Group 1 (UCMSCs - 20 million); Pilot Phase: Group 3 (UCMSCs - 100 million)
Biological: BMMSCs — Bone Marrow derived Mesenchymal Stem Cells (BMMSCs)
  Arms: Group B (BMMSCs - 100 million); Pilot Phase: Group 2 (BMMSCs - 20 million); Pilot Phase: Group 4 (BMMSCs -100 million)
Other: Placebo — a single administration of placebo delivered via peripheral intravenous infusion.
  Arms: Group C (Placebo)

SUMMARY:
This study is to compare the safety and efficacy of UCMSCs and BMMSCs administered intravenously in patients to evaluate cytokine suppression in patients with chronic inflammation. Cells administered via intravenous infusion (IV) and will be tested in 37 patients in two phases (Pilot and Randomized).

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Subjects age > 21 and < 95 years at the time of signing the Informed Consent Form.
* Each subject must have endothelial dysfunction.

Endothelial dysfunction Criteria:

Impaired flow-mediated vasodilation (FMD <7%)

• At the time of enrollment, each subject must meet at least 3 out of the 5 criteria under the harmonized definition of the metabolic syndrome, consisting of the following:

* Waist circumference - US defined: ≥ 102 cm (males) or ≥ 88 cm (females)
* Elevated triglycerides - ≥ 150 mg/dL (1.7 mM)
* Reduced HDL-C - Males: <40 mg/dL (1.0 mM) Females: <50 mg/dL (1.3 mM)
* Elevated blood pressure - Systolic ≥ 130 mm Hg and/or Diastolic ≥ 85 mm Hg
* Elevated fasting glucose - ≥ 100 mg/dL

Exclusion Criteria:

* Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods. Female subjects must undergo a blood or urine pregnancy test at screening and within 36 hours prior to infusion.
* Inability to perform any of the assessments required for endpoint analysis.
* Active listing (or expected future listing) for transplant of any organ.
* Clinically important abnormal screening laboratory values, as determined by the P.I.
* Serious comorbid illness or any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study.
* Have known allergies to penicillin or streptomycin.
* Hypersensitivity to dimethyl sulfoxide (DMSO).
* Be a solid organ transplant recipient. This does not include prior cell-based therapy (>12 months prior enrollment) bone, skin, ligament, tendon or corneal grafting. Have a history of organ or cell transplant rejection.
* Have a clinical history of malignancy within 3 years (i.e., subjects with prior malignancy must be disease free for 3 years), except curatively- treated basal cell carcinoma, squamous cell carcinoma, melanoma in situ or cervical carcinoma, if recurrence occurs.
* Have a non-pulmonary condition that limits lifespan to < 1 year.
* History of drug abuse (illegal "street" drugs except marijuana, or prescription medications not being used appropriately for a pre-existing medical condition) or alcohol abuse (≥ 5 drinks/day for ˃ 3 months), or documented medical, occupational, or legal problems arising from the use of alcohol or drugs within the past 24 months.
* Be serum positive for HIV, hepatitis B surface antigen or Viremic hepatitis C, and/or Syphilis.
* Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.
* Patients with Ejection Fraction <45% (heart failure patients).
* Glomerular Filtration Rate < or equal to 35 (chronic kidney disease stage 3 or higher).
* Liver disease (elevated Liver Function Tests greater than 3x normal limit).
* Advanced pulmonary disease (requiring home oxygen and/or less than 1 expected life span).
* Proliferative diabetic retinopathy
* Hemoglobin A1C greater than 7.

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2021-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Hare, MD, Principal Investigator — ISCI / University of Miami Miller School of Medicine
Locations (1):
- ISCI / University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Interdisciplinary Stem Cell Institute at the University of Miami Miller School website — http://isci.med.miami.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No subjects had been randomized to Group A or C at the time of trial termination.
Groups:
- Pilot Phase: Group 1 (UCMSCs - 20 Million): Three (3) subjects will be treated with a single administration of 2 x 10^7 (20 million) UCMSCs delivered via peripheral intravenous infusion.
  UCMSCs: Allogeneic Umbilical Cord Tissue derived Mesenchymal Stem Cells (MSC).
Period: Overall Study
Arm/Group | Pilot Phase: Group 1 (UCMSCs - 20 Million) | Pilot Phase: Group 2 (BMMSCs - 20 Million) | Pilot Phase: Group 3 (UCMSCs - 100 Million) | Pilot Phase: Group 4 (BMMSCs -100 Million) | Group A (UCMSCs - 100 Million) | Group B (BMMSCs - 100 Million) | Group C (Placebo)
Started | 3 | 3 | 3 | 3 | 0 | 2 | 0
Completed | 3 | 3 | 3 | 3 | 0 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized phase of the study was terminated after only 2 participants. No subjects were allocated to Group A or Group C in the randomized phase of the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Phase: Group 1 (UCMSCs - 20 Million) | Pilot Phase: Group 2 (BMMSCs - 20 Million) | Pilot Phase: Group 3 (UCMSCs - 100 Million) | Pilot Phase: Group 4 (BMMSCs -100 Million) | Group A (UCMSCs - 100 Million) | Group B (BMMSCs - 100 Million) | Group C (Placebo) | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 0 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 85.67 (5.13) | 62.00 (8.72) | 61.67 (12.9) | 60.67 (12.42) |  | 52 (12.73) |  | 65.17 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3
  Male | 2 | 2 | 3 | 2 | 0 | 2 | 0 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 5
  Not Hispanic or Latino | 3 | 2 | 2 | 1 | 0 | 1 | 0 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 2 | 3 | 3 | 2 | 0 | 1 | 0 | 11
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Serious Adverse Events (TE-SAEs)
Description: Number of treatment-emergent serious adverse events (SAE) (at one-month post infusion), defined as the composite of: death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities, determined per the Investigator's judgment.
Time Frame: one month post infusion
Population: No subjects had been randomized to Group A or C at the time of trial termination.
Measure: Number; unit: Events
Arm/Group | Pilot Phase: Group 1 (UCMSCs - 20 Million) | Pilot Phase: Group 2 (BMMSCs - 20 Million) | Pilot Phase: Group 3 (UCMSCs - 100 Million) | Pilot Phase: Group 4 (BMMSCs -100 Million) | Group A (UCMSCs - 100 Million) | Group B (BMMSCs - 100 Million) | Group C (Placebo)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 0
Events | 0 | 0 | 0 | 0 |  | 0 |

2. Secondary Outcome: Cytokine Levels
Description: Cytokine levels including the following panel of inflammatory and angiogenic markers: Interleukin-1 (IL-1), Interleukin-6 (IL-6), Tumor Necrosis Factor alpha (TNFα), and Vascular Endothelial Growth Factor (VEGF), & Stromal Cell Derived Factor (SDF-1a) levels from serum/plasma samples all measured in pg/mL.
Time Frame: at Baseline, at Week 2, at Month 1, at Month 3, and at Month 6
Population: Some participants did not complete all of the study visits per protocol due to COVID-19 pandemic restrictions. Therefore not all data is available for all time-points for all participants.
  Blood samples were collected for IL-1 and SDF-1a analysis, however due to cost and logistical reasons the samples were not analyzed.
  VEGF were to be analyzed internally using frozen plasma aliquots. No plasma samples were retained for internal testing at week 2, month 1, and month 6 in all participants.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pilot Phase: Group 1 (UCMSCs - 20 Million) | Pilot Phase: Group 2 (BMMSCs - 20 Million) | Pilot Phase: Group 3 (UCMSCs - 100 Million) | Pilot Phase: Group 4 (BMMSCs -100 Million) | Group A (UCMSCs - 100 Million) | Group B (BMMSCs - 100 Million) | Group C (Placebo)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 0
pg/mL
  IL-6 Baseline | 5.7 (4.8) | 2.7 (1.8) | 3.2 (2.5) | 2.9 (1.9) |  | 1.2 (0.6) |
  IL-6 Week 2 | 5.8 (5.2) | 3.4 (1.0) | 5.4 (6.7) | 3.7 (2.3) |  | 1.4 (0.4) |
  IL-6 Month 1: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 1 | 0
  IL-6 Month 1 | 5.4 (3.9) | 2.8 (1.0) | 2.5 (1.0) | 2.1 (0.9) |  | 1.3 |
  IL-6 Month 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0
  IL-6 Month 3 | 8.4 (4.5) | 2.5 (1.2) | 1.9 (0.6) | 2.3 (1.0) |  |  |
  IL-6 Month 6: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 0 | 0
  IL-6 Month 6 | 2.9 (2.2) | 3.2 (1.3) | 3.8 (3.0) | 2.2 (0.4) |  |  |
  TNFa Baseline | 1.7 (0.4) | 1.6 (0.4) | 1.6 (0.8) | 2.1 (0.5) |  | 1.1 (0.2) |
  TNFa Week 2: number analyzed (Participants) | 3 | 2 | 3 | 3 | 0 | 2 | 0
  TNFa Week 2 | 1.9 (0.8) | 1.5 (0.6) | 1.5 (0.6) | 2.1 (0.7) |  | 0.9 (0.3) |
  TNFa Month 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 1 | 0
  TNFa Month 1 | 1.7 (1.1) | 1.5 (0.3) | 2.0 (0.9) | 2.2 (0.8) |  | 0.7 |
  TNFa Month 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 1 | 0
  TNFa Month 3 | 2.2 (1.7) | 1.2 (0.5) | 1.8 (1.0) | 1.8 (0.5) |  | 0.7 |
  TNFa Month 6: number analyzed (Participants) | 3 | 3 | 3 | 2 | 0 | 1 | 0
  TNFa Month 6 | 1.5 (0.6) | 1.4 (0.3) | 1.4 (0.3) | 1.0 (0.5) |  | 0.5 |
  VEGF Baseline: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0
  VEGF Baseline | 13.5 (4.8) | 19.2 (9) | 25.1 (14) | 13.5 (1.7) |  |  |
  VEGF Month 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0
  VEGF Month 3 | 15.3 (3) | 16.5 (12.4) | 15.5 (6.4) | 9.5 (1.8) |  |  |

3. Secondary Outcome: hsCRP Levels
Description: values at baseline and follow up for the following inflammatory marker: Serum High sensitivity C-Reactive Protein (hsCRP) in mg/L.
Time Frame: at Baseline, at Week 2, at Month 1, at Month 3, and at Month 6
Population: No subjects had been randomized to Group A or C at the time of trial termination. Some participants did not complete all of the study visits per protocol.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pilot Phase: Group 1 (UCMSCs - 20 Million) | Pilot Phase: Group 2 (BMMSCs - 20 Million) | Pilot Phase: Group 3 (UCMSCs - 100 Million) | Pilot Phase: Group 4 (BMMSCs -100 Million) | Group A (UCMSCs - 100 Million) | Group B (BMMSCs - 100 Million) | Group C (Placebo)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 0
mg/L
  Baseline | 2.0 (1.6) | 13.0 (19.2) | 1.4 (0.4) | 3.2 (1.9) |  | 0.5 (0.3) |
  Week 2 | 9.2 (14.4) | 5.7 (6.0) | 1.7 (1.4) | 4.3 (3.3) |  | 0.6 (0.3) |
  Month 1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 1 | 0
  Month 1 | 10.7 (16.0) | 4.6 (4.0) | 2.1 (1.4) | 2.9 (1.2) |  | 0.6 |
  Month 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 1 | 0
  Month 3 | 5.0 (3.4) | 4.7 (5.1) | 2.7 (2.9) | 3.4 (1.3) |  | 0.9 |
  Month 6: number analyzed (Participants) | 2 | 3 | 2 | 1 | 0 | 1 | 0
  Month 6 | 1.6 (1.1) | 5.4 (7.0) | 2.6 (1.2) | 2.1 |  | 0.6 |

4. Secondary Outcome: Stem Cell Factor (SCF) Levels
Description: SCF levels from serum/plasma samples measured in units of mg/mL
Time Frame: at Baseline, at Week 2, at Month 1, at Month 3, and at Month 6
Population: Blood samples were collected for SCF analysis, however due to cost and logistical reasons the samples were not analyzed and hence no data were generated.
Arm/Group | Pilot Phase: Group 1 (UCMSCs - 20 Million) | Pilot Phase: Group 3 (UCMSCs - 100 Million) | Pilot Phase: Group 2 (BMMSCs - 20 Million) | Pilot Phase: Group 4 (BMMSCs -100 Million) | Group A (UCMSCs - 100 Million) | Group B (BMMSCs - 100 Million) | Group C (Placebo)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Endothelial Progenitor Cell-Colony Forming Units (EPC-CFUs)
Description: Endothelial function will be reported as the change in Endothelial Progenitor Cell Colony Forming Unit (EPC-CFU) assessed via blood sample assay
Time Frame: at Baseline, and at 3 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Colony Forming Units per Well
Arm/Group | Pilot Phase: Group 1 (UCMSCs - 20 Million) | Pilot Phase: Group 2 (BMMSCs - 20 Million) | Pilot Phase: Group 3 (UCMSCs - 100 Million) | Pilot Phase: Group 4 (BMMSCs -100 Million) | Group A (UCMSCs - 100 Million) | Group B (BMMSCs - 100 Million) | Group C (Placebo)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 0
Colony Forming Units per Well
  Baseline | 15.0 (14.5) | 0.8 (0.9) | 2.3 (3.1) | 4.8 (6.6) |  | 0.6 (0.6) |
  Month 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0
  Month 3 | 20.4 (20.8) | 1.3 (1.1) | 13.2 (13.6) | 1.9 (2.0) |  |  |

6. Secondary Outcome: Flow Mediated Diameter Percentage (FMD%)
Description: FMD% will be assessed using brachial artery ultrasound
Time Frame: at Baseline and at Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of change in brachial artery
Arm/Group | Pilot Phase: Group 1 (UCMSCs - 20 Million) | Pilot Phase: Group 2 (BMMSCs - 20 Million) | Pilot Phase: Group 3 (UCMSCs - 100 Million) | Pilot Phase: Group 4 (BMMSCs -100 Million) | Group A (UCMSCs - 100 Million) | Group B (BMMSCs - 100 Million) | Group C (Placebo)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 2 | 0
percentage of change in brachial artery
  Baseline | 3.6 (2.0) | 4.1 (1.1) | 3.6 (0.8) | 3.1 (1.4) |  | 5.0 (0.8) |
  Month 3: number analyzed (Participants) | 3 | 3 | 3 | 3 | 0 | 0 | 0
  Month 3 | 3.5 (1.9) | 5.4 (3.7) | 5.4 (0.5) | 4.0 (0.8) |  |  |

ADVERSE EVENTS:
Time Frame: 1 year
Description: No subjects had been randomized to Group A or C at the time of trial termination.
Arm/Group | Pilot Phase: Group 1 (UCMSCs - 20 Million) | Pilot Phase: Group 2 (BMMSCs - 20 Million) | Pilot Phase: Group 3 (UCMSCs - 100 Million) | Pilot Phase: Group 4 (BMMSCs -100 Million) | Group A (UCMSCs - 100 Million) | Group B (BMMSCs - 100 Million) | Group C (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/0 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 0/3 | 0/3 | 0/0 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 2/3 | 3/3 | 0/0 | 1/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Phase: Group 1 (UCMSCs - 20 Million) (N=3) | Pilot Phase: Group 2 (BMMSCs - 20 Million) (N=3) | Pilot Phase: Group 3 (UCMSCs - 100 Million) (N=3) | Pilot Phase: Group 4 (BMMSCs -100 Million) (N=3) | Group A (UCMSCs - 100 Million) (N=0) | Group B (BMMSCs - 100 Million) (N=2) | Group C (Placebo) (N=0)
Esophageal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot Phase: Group 1 (UCMSCs - 20 Million) (N=3) | Pilot Phase: Group 2 (BMMSCs - 20 Million) (N=3) | Pilot Phase: Group 3 (UCMSCs - 100 Million) (N=3) | Pilot Phase: Group 4 (BMMSCs -100 Million) (N=3) | Group A (UCMSCs - 100 Million) (N=0) | Group B (BMMSCs - 100 Million) (N=2) | Group C (Placebo) (N=0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monoclonal Gammopathy of Uncertain Significance (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congestive Heart Falure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital Hematoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes Mellitus Type 2 (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 3 (3) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injured Ankle (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toenail Avulsion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toe Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine Elevation (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver Enzyme Elevation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left Foot Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lump on Elbow (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RIght Leg Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rupture of Left Distal Biceps Tendon (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vocal Cord Paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasovagal Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migrane Exacerbation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Microhematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic Left Foot Ulcers (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scalp Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral Vascular Disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudoaneurysm of Right Femoral Artery (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated Blood Pressure (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left Arm Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Funding timeline was not met due to the coronavirus disease 2019 (COVID-19) pandemic. No additional funding was provided, therefore the study had to be terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03059355/Prot_SAP_000.pdf